CLINICAL TRIAL: NCT06732765
Title: Comparative Effects of Eldoa With and Without Muscle Energy Technique on Pain, Range of Motion and Functional Disability in Patient With Quadratus Lumborum Syndrome
Brief Title: Comparative Effects of Eloda With/Without Muscle Energy Technique in Patient With Quadratus Lumborum Syndrome
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: REC/RCR&AHS/24/0123
Record Dates: First submitted 2024-11-25; First posted 2024-12-13 (Actual); Last update posted 2024-12-13 (Actual); Status verified 2024-12

CONDITIONS: Rounded Shoulder Posture

STUDY DESIGN:
Who Masked: Participant, Investigator
Masking Description: The Study will be single blind, assessor will be kept blind because patients and clinicians were difficult to mask due to well distinguished treatment protocol.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Pilates exercise program (Experimental): Pilates exercise program Will be treated with WBV with Pilate Exercises. Before applying exercise, hot pack will be applied for 15-20minutes
  Interventions: Other: Pilates exercise program
- Traditional physical therapy program (Active Comparator): traditional physical therapy program in form of stretching, strengthening and postural correction exercises
  Interventions: Other: Traditional physical therapy program

INTERVENTIONS:
Other: Pilates exercise program — Pilates exercise program Will be treated with WBV with Pilate Exercises. Before applying exercise, hot pack will be applied for 15-20minutes
  Arms: Pilates exercise program
Other: Traditional physical therapy program — Traditional physical therapy program in form of stretching, strengthening and postural correction exercises
  Arms: Traditional physical therapy program

SUMMARY:
The aim of the study is to compare effects Comparison of Pilate exercises with and without whole body vibration on posture, disability and pain in patients with upper cross syndrome. A randomized contro ltrial will beconductedat PESSI. Non-probability convenience sampling will be used, and 62 subjects, age 20-40 years will be allocated into two groupsby the computer generated software after meeting the inclusion criteria. Both groups will receive hot pack for 15-20 minutes and Pilate exercises perform both groups as common treatment.Group A will be treated with Pilate exercisesandGroupB will be treated with Pilate exercise with whole body vibration both groups received two sessions per week for four consecutive weeks by another well trained physical therapist. Session duration for both groups ranged from 55 minutes to 1 hour. 2 sessions for 4 weeks will be given. The outcome measures will be conducted through NPRS, NDI, RSP WAS MEASURED IN SUPINE POSITION AND THEN PML AND TSD and J APP/ software before and after 4 weeks. Data will be analyzed using SPSS software version 26.After assessing normality of data by kolmo-grove test, it will be decided either parametric or non-parametric test will be used within a group or between two groups. Data will be collected at baseline and after 4 weeks of follow up.

DETAILED DESCRIPTION:
In 2023, conducted the study in Basic Science Department,. Forty participants (females) with UCS were randomly divided into two equal groups: group A (control group) and group B (experimental group). Both groups received two sessions per week for four consecutive weeks. Group A received traditional physical therapy program in form of stretching, strengthening and postural correction exercises while Group B received Pilates exercise program. Primary outcome measures were balance, spinal curvature, Craniovertebral angle (CV), and rounded shoulders. Result was Comparison between pre-and post-treatment .Conclusions was Pilates exercise program proved better than traditional physical therapy program in improving spinal curvature, balance, and function and reducing pain in UCS.Randomized clinical trials (RCTs) were conducted to identify the effectiveness of whole-body vibration (WBV) on strength, power, and muscular endurance in older adults. However, the results of different studies are contradictory.. Conclusion: WBV was effective in increasing lower limb muscle strength. However, no significant results were observed for upper limb strength, lower limb power, and lower and upper limb muscle endurance in older adults. However, more studies are needed to better understand the physiological impacts of WBV in older.A randomized controlled trial was conducted in 2017.The present study aimed to determine the immediate effects of Whole Body vibration (WBV) on Rounded Shoulder Posture (RSP) in healthy women. Thirty female students aged between 18 to 30 years with RSP participated in this study. First, the examiner measured the RSP (in supine position), Pectoralis Minor Length (PML) and Total Scapular Distance (TSD). Then, the subjects performed 5 sets of 1-min WBV (frequency=30 Hz, amplitude=5 mm) with 1 min rest between each set. After intervention, the examiner immediately measured the above mentioned variables. The paired t test was used for data analysis. The analysis showed that WBV significantly decreased the supine measurement of RSP (P<0.001) and TSD (P=0.03) and increased PML (P <0.001). It seems that WBV had immediate effect on postural correction of rounded shoulder posture in the study subjects.While posture is a prevalent issue among young adults due to prolonged sitting and increase use oftechnology, the majorityofresearch studies have primarily focused on other age groups, such as older adults or adolescents and most of work on lower limb , very little study was done in upper limb regarding this issue among young adults.As my study focus posture correction in upper croos syndrom patient . After study some literature found to the best of authors knowledge, although in the past many studies have worked on correction ofposture leading to forward head posture and rounded shoulder in upper cross syndrome.There are different exercise regimes for RSP such as strengthening of lengthened muscles, scapular stabilizers, stretching of shorten muscles especially pectoral muscles, and soft tissue mobilization Pilate exercises and whole body vibration have been practiced in the treatment of forward head posture and RSP were found effective individually,butthereisalackofComparison of pilot exercises with and without whole body vibration on posture , disability and pain in patients with upper cross syndrome . This RCT aims to evaluate the effect of WBV with exercise and effect of Pilate exercises without WBV will ascertain thatiftwoofthese mayhave differenteffectsonthepain, posture, disability in young adults with upper cross syndrome.

ELIGIBILITY:
Inclusion Criteria:

* Age group between 18 to 45 years
* Both gender male and female
* individuals with mechanical lower back pain
* active trigger point in the quadratus lumborum muscle
* No previous history of accidents

Exclusion Criteria:

* Acute muscular injuries
* localized or systemic infections
* lumbar disc herniation
* spinal abnormalities, any prior history of spinal
* anticoagulant use and bleeding disorders
* psychiatric conditions that would have made it difficult to provide consent

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 62 (Estimated)
Dates: Start 2024-02-04 (Actual); Primary Completion 2024-12-07 (Estimated); Study Completion 2025-01-15 (Estimated)

PRIMARY OUTCOMES:
Numeric Pain Rating Scale (NPRS) | 6 weeks
  The Numeric Pain Rating Scale (NPRS) (an outcome measure) that is a unidimensional measure of pain intensity in adults,Numeric Pain Rating Scale (NRS-11), which is an eleven-point scale in which the end points are the extremes of no pain at all (score of 0) and the worst pain the patient has ever experienced (score of 10)
Universal Goniometer (UG) | 6 weeks
  Universal Goniometer (UG) The measurement of joint range of motion (ROM) is an essential procedure used in physical therapy, known as goniometry[24].Goniometry, the measurement of joint angles, traditionally performed with a universal goniometer (UG), is a commonly utilized assessment tool in monitoring problems of the musculoskeletal system, as well as the progression of rehabilitation interventions
Modified Oswestry Disability Index (MODI) | 6 weeks
  The Oswestry Disability Index (ODI) a patient-completed questionnaire .It provides patients receiving low back pain rehabilitation with a subjective percentage score of their degree of function (disability) in everyday activities. it has become one of the most widely used outcome measures for low back pain

CONTACTS AND LOCATIONS:
Overall Officials: Muhammad Salman, PhD, Principal Investigator — Riphah International University
Locations (1):
- Muhammad Sulman, Sialkot, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No